CLINICAL TRIAL: NCT07066930
Title: Optimizing Alveolar Ridge Expansion: A Clinical Comparison of Magneto-Dynamic Ridge Splitting and Versah Osseodensification Techniques
Brief Title: Optimizing Alveolar Ridge Expansion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Collaborators: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Abduljaleel Azad Koyi, Optimizing Alveolar Ridge Expansion: A Clinical Comparison of Magneto-Dynamic Ridge Splitting and Versah Osseodensification Techniques, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMUD2425177
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Dental Implant
Keywords: Ridge expansion; Osseodensification; Magnetic mallet; Dental implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magneto-Dynamic Ridge Splitting (Experimental): Participants in this arm will undergo ridge expansion using the Magnetic Mallet system. The procedure involves magneto-dynamic impulses to laterally expand the alveolar ridge prior to dental implant placement.
  Interventions: Procedure: Magneto-Dynamic Ridge Expansion
- Versah Osseodensification (Active Comparator): Participants in this arm will undergo ridge expansion using Versah drills (Densah burs) in osseodensification mode prior to dental implant placement.
  Interventions: Procedure: Osseodensification with Versah Drills

INTERVENTIONS:
Procedure: Magneto-Dynamic Ridge Expansion — A ridge expansion technique using the Magnetic Mallet device. Controlled magneto-dynamic impulses are applied to split the alveolar ridge and compact bone prior to immediate implant placement.
  Arms: Magneto-Dynamic Ridge Splitting
Procedure: Osseodensification with Versah Drills — A ridge expansion method using Versah drills (Densah burs) in osseodensification mode. The drills densify bone without removing it, enhancing bone density and implant stability.
  Arm Assignment: Versah Osseodensification (Active Comparator arm)
  Arms: Versah Osseodensification

SUMMARY:
The goal of this clinical trial is to compare two surgical techniques-Magneto-Dynamic Ridge Splitting and Versah Osseodensification-for expanding narrow alveolar ridges in adults requiring dental implant placement. The main questions it aims to answer are:

Which technique better preserves alveolar bone width after surgery?

Which method results in higher primary implant stability?

Researchers will compare ridge splitting using the Magnetic Mallet to ridge expansion using Versah drills to see if one technique leads to better clinical outcomes, such as improved bone preservation, greater implant stability, and favorable soft tissue response.

Participants will:

Undergo ridge expansion surgery using either the Magnetic Mallet or Versah drills, followed by immediate dental implant placement.

Receive CBCT scans before and 4 months after surgery to measure bone changes.

Undergo implant stability testing using the ISQ (Implant Stability Quotient) method.

Have intraoral scans to evaluate changes in soft tissue volume and thickness.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate and compare two innovative techniques used to widen narrow jawbone areas (alveolar ridges) in preparation for dental implants. In many patients, the bone in the jaw may be too thin to support dental implants without additional procedures. Traditionally, this problem has been addressed using more invasive surgical methods that can involve bone grafting and extended healing times.

The two techniques being studied are:

Magneto-Dynamic Ridge Splitting (Magnetic Mallet) - This method uses gentle electromagnetic impulses to gradually split and expand the bone. The technique is minimally traumatic, preserves the outer bone layer (cortical bone), and may promote better healing and stability for implants.

Osseodensification (Versah Drills) - This technique uses specially designed rotating drills (Densah burs) that do not remove bone but instead compact it outward, increasing its density. This approach is designed to strengthen the implant site and improve how well the implant integrates with the bone.

The study is a randomized controlled clinical trial conducted at Hawler Medical University. Participants will be randomly assigned to one of the two groups. Both groups will receive immediate implant placement following the ridge expansion procedure, using the same implant system (ROOTT Implants).

Key outcomes to be measured include:

Changes in bone width (buccolingual ridge dimension) using Cone Beam Computed Tomography (CBCT) before and 4 months after surgery.

Implant Stability Quotient (ISQ) values recorded at the time of implant placement and again during the second-stage surgery using a non-invasive resonance frequency analysis device (Osstell).

Soft tissue changes, such as thickness and volume around the implant site, using intraoral scanning technology.

The trial will also monitor patient comfort, healing, and potential complications in each group. By directly comparing these two methods, the researchers hope to determine which approach provides better clinical outcomes in terms of bone preservation, implant stability, and soft tissue health. The results may help establish a new standard in minimally invasive implant site preparation techniques and guide oral surgeons and implantologists in choosing the most effective ridge expansion strategy for their patients.

This study will be conducted in accordance with ethical standards, and all participants will be asked to provide informed consent prior to joining the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years.
* Partially edentulous patients requiring ridge expansion prior to dental implant placement.
* Alveolar ridge width between 4 mm and 6 mm as measured on CBCT.
* Sufficient vertical bone height for implant placement without the need for vertical augmentation.
* Adequate oral hygiene and commitment to postoperative care and follow-up visits.
* Signed informed consent form.

Exclusion Criteria:

* Presence of systemic conditions contraindicating oral surgery (e.g., uncontrolled diabetes, immune-compromised status).
* History of bisphosphonate therapy or radiation therapy to the head and neck region.
* Active periodontal disease or untreated oral infections.
* Heavy smokers (more than 10 cigarettes per day).
* Pregnant or breastfeeding women.
* History of substance abuse or psychiatric disorders that could impair compliance with study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Alveolar Ridge Width (Buccolingual Dimension) | 4 Months
  Measurement of alveolar ridge width in millimeters using Cone Beam Computed Tomography (CBCT) to assess the horizontal bone gain after ridge expansion with either the Magneto-Dynamic Ridge Splitting or Versah Osseodensification technique.
Change in Alveolar Ridge Width (Buccolingual Dimension) | Baseline (pre-operative) and 4 months post-surgery
  Measurement of alveolar ridge width in millimeters using Cone Beam Computed Tomography (CBCT) to assess the horizontal bone gain after ridge expansion with either the Magneto-Dynamic Ridge Splitting or Versah Osseodensification technique.

CONTACTS AND LOCATIONS:
Overall Officials: Jodal Ahmed, PhD, Study Director — Oral and Maxillofacial Surgery Department, College of Dentistry, Hawler Medical University, Erbil, Kurdistan Region, Iraq.
Locations (1):
- Oral and Maxillofacial Surgery Department, College of Dentistry, Hawler Medical University, Erbil, Kurdistan Region, Iraq., Erbil, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet determined whether individual participant data (IPD) will be shared with other researchers. The decision will depend on the outcomes of the study, institutional policies, ethical approvals, and potential publication requirements. Any future data sharing will comply with applicable data protection regulations and will require appropriate de-identification and ethical clearance.

REFERENCES:
- See also: Related Info — https://www.osseotouch.com/en/magnetic-mallet/
- See also: Related Info — https://versah.com/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT07066930/Prot_SAP_ICF_000.pdf